CLINICAL TRIAL: NCT00511056
Title: Adherence and Risk Behaviour in Patients With HIV Infection Receiving Antiretroviral Therapy
Acronym: ARB
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT Amendment II to 006
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: HIV; Adherence; Compliance; Highly Active Antiretroviral Therapy (HAART); ARV; ART; Sexual Risk Behavior; Unsafe; Transmission
MeSH Terms: conditions — HIV Infections; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples required to provide Viral Load data and CD4 cell count
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIVNAT 006: HIVNAT 006 is a long term follow up cohort. The primary objective of this study is to collect and evaluate the long-term clinical outcomes of HIV infected patients have participated in HIV-NAT studies. These subjects will be used to test our hypothesis.

SUMMARY:
Study Hypothesis: Do certain risk behaviours impact/predict levels of HIV antiretroviral adherence?

Objectives:

* To assess risk behavior in HIV-positive individuals receiving highly active antiretroviral therapy.(HAART)
* To assess levels of adherence in the same subjects at the same time point
* To determine if there is a correlation between HAART adherence and risk behaviour

DETAILED DESCRIPTION:
Background and Rationale:

Adherence to an effective antiretroviral (ARV) regimen is the most important determinant of treatment success in patients receiving ARV. It is now well established that virological suppression on highly active antiretroviral therapy (HAART) requires strict adherence to prescribed dosing schedules. It is essential to reach and maintain therapeutic levels of these drugs, and strict adherence is particularly crucial for preventing the development of drug-resistant viral strains. If therapeutic drugs levels are suboptimal and the virus is able to replicate, this has important individual and public health implications.

Indirect evidence also suggests that the use of HAART by HIV-infected individuals decreases sexual transmission of HIV. Specifically, ARV treatment decreases serum and genital fluid HIV viral load. It has become evident that the availability of HAART may paradoxically increase sexual practices that lead to HIV transmission. This has been seen in several developed countries where the introduction of HAART coincided with increasing sexual risk behaviour and sexually transmitted infections. Thus far there has been very little evidence showing these trends in developing countries.

Despite the high burden on HIV in developing countries compared with developed countries, considerably more evidence is available in the latter regarding adherence and risk behaviour. Studies to ascertain the correlation between these two factors are important as new interventions may be established to ensure that improved health and economic outcomes will follow. Understanding which patients have increased risk behaviours, or are at risk for non-adherence enables identification of patients who are important targets for interventional strategies to optimise HIV treatment programmes.

Adherence and risk behaviour:

Apart from the beneficial clinical effects of HAART, treatment advances may have unintended effects on sexual behaviour. Evidence suggests that since HAART became available, the prevalence of unprotected sex and the incidence of sexually transmitted infections including HIV have increased, mostly among men who have sex with men (MSM). Some HIV positive persons receiving HAART, especially those with a undetectable viral load, may feel protected from transmitting HIV sexually. Recent evidence does suggest that an undetectable viral load may reduce the level of infectiousness of HIV positive persons receiving HAART.

As this information moves into the public domain it may influence peoples beliefs about HIV transmission and lessen concern about engaging in unsafe sex. People who hold these beliefs are more likely than their counterparts to engage in unprotected sex.

HIV positive patients who engage in high-risk behaviours linked to HIV spread are as likely to be receiving HAART as those at low risk for disease transmission, but those who engage in high-risk behaviours have much lower rates of medication adherence and thus much higher viral loads. This suggests a strong behavioural basis for transmission of drug resistant HIV, and parallels recent increases in all sexually transmitted infections. Given that taking HAART and having an undetectable viral load do not eliminate the possibility of transmitting HIV, it is important to examine whether the use of HAART and beliefs about HAART are associated with sexual risk taking.

Definitions:

Risk behavior is defined as behavior which may result in transmission of HIV

Study subjects:

Subjects will be asked to complete a questionnaire which will contain questions on adherence and risk behaviour.At the completion of data collection an analysis will be made accordingly. Approximately 700 patients in HIV-NAT 006 who provide consent will be enrolled.

Inclusion criteria are:

* Age ≥ 18 years
* HIV seropositive.
* On continuous HAART for at least 6 months
* Signed written informed consent

Methods:

Cross sectional survey of adherence and behavior in subjects enrolled in the HIVNAT 006 long term follow up cohort.

Patients enrolled in HIVNAT 006 are normally required to attend regular 6 monthly follow up appointments. Over the coming months 700 subjects who give consent will be asked to complete an anonymous self-administered questionnaire at their next clinic visit. Completion of the questionnaire will be facilitated by people living with HIV/AIDS (PLHA) who will be trained by HIVNAT.

The questionnaire will comprise the following categories:

1. Demographics
2. Medication adherence
3. Factors affecting adherence (risk behaviour)

Furthermore the following will be extracted from the HIVNAT database:

* CDC disease stage over the previous 12 months and at current consult
* CD4 over the previous 12 months and at current consult
* VL over the previous 12 months and at current consult
* ARV regimen and changes in regimen
* Opportunistic infections

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* HIV seropositive.
* On continuous HAART for at least 6 months
* Signed written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 500 subjects were surveyed from the HIVNAT 006 long term follow up cohort. A sample size as large as this is likely to yield accurate results as to the true relationship between sexual risk behavior and adherence to HIV medications.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The relationship between sexual risk behavior and adherence to HIV medications and how do these behaviors relate to patient beliefs about HIV transmission. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, M.D., M.Sc., Principal Investigator — HIVNAT
Locations (1):
- HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok, Thailand

REFERENCES:
- [Result] Honeybrook AL. Adherence and Risk Behaviour in Patients With HIV Recieving antiretroviral therapy. XVII International AIDS Conference 2008. Mexico City, Mexico.
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org